CLINICAL TRIAL: NCT00217672
Title: A Randomized Phase II Trial of Docetaxel With or Without Bevacizumab as First-Line Therapy for Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Metastatic Breast Cancer
Brief Title: Docetaxel With Bevacizumab as First-Line Therapy in Treating Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000442877; UCLA-0501049-01 (Other: UCLA); TORI-B-01 (Other: UCLA); NCT00203398 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab + Docetaxel (Experimental): docetaxel: 75 mg/m2 IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.
  Bevacizumab: 15 mg/kg IV every 3 weeks. Subjects continue on study until disease progression, unacceptable toxicity, or withdrawal of patient consent.
  Interventions: Biological: bevacizumab; Drug: Docetaxel
- docetaxel (Active Comparator): docetaxel: 75 mg/m2 IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: bevacizumab — Patients receive bevacizumab 15 mg/kg intravenously (I.V.) every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal.
  Arms: Bevacizumab + Docetaxel
Drug: Docetaxel — docetaxel: 75 mg/m2 IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by stopping blood flow to the tumor. It is not yet known whether giving docetaxel together with bevacizumab is more effective than docetaxel alone in treating breast cancer.

PURPOSE: This randomized phase II trial is studying how well giving docetaxel together with bevacizumab works compared to docetaxel alone as first-line therapy in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
This trial began as a 2-arm study with a docetaxel-alone arm. When bevacizumab became widely available, it was converted to a 1-arm open-label trial of docetaxel/bevacizumab. Patients enrolled in the docetaxel-alone arm were permitted to cross over to docetaxel/bevacizumab. Patients received bevacizumab 15 mg/kg and docetaxel 75 mg/m2 intravenously (I.V.) every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal.

ELIGIBILITY:
Inclusion Criteria

* Female 18 and over
* Histologically or cytologically confirmed adenocarcinoma of the breast at first diagnosis
* Stage IV disease, with at least one measurable lesion according to the RECIST criteria.
* HER2-negative disease, by fluorescence in situ hybridization
* ECOG performance status 0-1
* Life expectancy of at least 24 weeks
* No prior chemotherapy for metastatic breast cancer (prior endocrine therapy is permitted).
* Prior adjuvant chemotherapy is permitted. If patients received a taxane in the adjuvant setting, at least 12 months must have elapsed since the completion of adjuvant therapy.
* At least 4 weeks since prior surgery, radiotherapy, endocrine therapy, or experimental drug therapy, with complete recovery from the effects of these interventions
* If female of childbearing potential, pregnancy test is negative and willing to use effective contraception while on treatment for at least 3 months thereafter.
* Patient is accessible and willing to comply with treatment and follow-up.
* Patient is willing to provide written informed consent prior to the performance of any study-related procedures.
* Required laboratory values

  * Absolute neutrophil count ≥ 1,500/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Hemoglobin ≥ 9.0 g/dL
  * Creatinine ≤ 2.0 mg/dL
  * Total bilirubin < 1.0 x upper limit of normal (ULN) (patients with documents Gilbert's syndrome are eligible).
  * Alkaline phosphatase (AP) normal AND Angiotensin Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN) or AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN or AP ≤ 5 times ULN AND AST or ALT normal.

Exclusion Criteria

* Prior chemotherapy for metastatic breast cancer
* Prior treatment with an anti-angiogenic agent
* Concurrent therapy with any other non-protocol anti-cancer therapy
* Current or prior history of central nervous system or brain metastases
* Presence of neuropathy > grade 2 (NCI- Common Toxicity Criteria (CTC) version 3.0) at baseline
* Presence of any non-healing wound, fracture, or ulcer, or the presence of clinically significant (> grade 2) peripheral vascular disease
* History of any other malignancy within the past 5 years, with the exception of non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension [BP > 150/100]), myocardial infarction or stroke within the past 6 months, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* Active peptic ulcer disease, inflammatory bowel disease, or other gastrointestinal condition increasing the risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning therapy
* Active, uncontrolled infection requiring parenteral antimicrobials
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of the drugs in this protocol or place the subject at undue risk for treatment complications.
* Inability to comply with the study protocol or follow-up procedures
* Pregnancy or lactation
* A history of a severe hypersensitivity reaction to Bevacizumab, or Docetaxel or other drugs formulated with polysorbate 80.
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study; minor surgical procedure, fine needle aspiration or core biopsy within 7 days prior to beginning therapy
* Proteinuria at baseline or clinically significant impairment of renal function. Subjects unexpectedly discovered to have > 1+ proteinuria at baseline should undergo a 24 hour urine collection, which must be an adequate collection and must demonstrate <1 gm of protein/24 hour to allow participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hurvitz, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from March 2005 to September 2006 at academic medical clinics and community medical clinics.
Groups:
- Docetaxel+Bevacizumab: docetaxel: 75 mg/m2 IV q3 weeks. Bevacizumab: 15mg/kg IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.
Period: Allocation
Arm/Group | Docetaxel+Bevacizumab | Docetaxel
Started | 69 | 7 (When bevacizumab became available, study converted to a 1-arm open-label trial with just bevacizumab)
Completed | 67 | 7
Not Completed | 2 | 0
Not completed — Ineligible | 2 | 0
Period: Treatment
Arm/Group | Docetaxel+Bevacizumab | Docetaxel
Started | 67 | 7 (When bevacizumab became available, study converted to a 1-arm open-label trial with just bevacizumab)
Completed | 0 | 0
Not Completed | 67 | 7
Not completed — disease progression | 33 | 4
Not completed — Adverse Event | 18 | 2
Not completed — reqd treatment not permitted by protocol | 6 | 0
Not completed — Physician Decision | 6 | 0
Not completed — insurance issues | 1 | 1
Not completed — Death | 2 | 0
Not completed — secondary malignancy | 1 | 0
Period: Follow-up
Arm/Group | Docetaxel+Bevacizumab | Docetaxel
Started | 74 (when bevacizumab became available, converted to a 1-arm open-label trial (67+7=74)) | 0
Completed | 69 | 0
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel + Bevacizumab: docetaxel: 75 mg/m2 IV q3 weeks. Bevacizumab: 15mg/kg IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.
  A total of 104 participants were screened for the study. Twenty six participants did not meet eligibility criteria and 2 withdrew consent.
  Seventy six participants were registered to the Treatment Period, 7 to arm A and 69 to arm B. Six out of 7 participants randomized to arm A elected to cross over to arm B once bevacizumab became available. Two out of the 69 participants randomized to arm B were found ineligible and taken off study before receiving treatment. As a result, the efficacy analysis was performed on 67 patients.
Arm/Group | Docetaxel + Bevacizumab
Number analyzed (Participants) | 67
Age, Continuous [Median (Full Range); unit: years] | 57 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 46
  More than one race | 0
  Unknown or Not Reported | 8
Hormone receptor status [Number; unit: participants]
  Estrogen Receptor(ER)+ Progesterone Receptor(PR)+ | 29
  ER+PR- | 13
  ER-PR+ | 3
  ER-PR- | 22
Number of metastatic sites [Number; unit: participants]
  less than 3 | 37
  more than 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity Based on Time to Tumor Progression (TTP).
Time Frame: From randomization until tumor progression
Population: 76 participants were registered to the Treatment, 7 to arm A and 69 to arm B. 6 participants randomized to arm A elected to cross over to arm B once Avastin became available. 2 out of the 69 participants randomized to arm B were found ineligible and taken off study before receiving treatment. Thus, the efficacy analysis performed on 67 patients.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Docetaxel + Bevacizumab: docetaxel: 75 mg/m2 IV q3 weeks. Bevacizumab: 15mg/kg IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.
Arm/Group | Docetaxel + Bevacizumab
Number analyzed (Participants) | 67
months | 9.3 [8.2 to 12.4]

2. Secondary Outcome: Comparison of Response Rates, Duration of Response, and Overall Survival
Time Frame: Time of death, up to 3 years
Population: Response rate - the percentage of patients assigned to a treatment arm who experience a CR or PR. Duration of response - the interval from date of initial documented response (CR or PR) to the first documented date of disease progression. Overall survival - the interval from the date of registration and the date of death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel + Bevacizumab
Number analyzed (Participants) | 67
months
  Overall Duration of Response (DR) | 11.8 [9.0 to 18.2]
  Overall Observed Response (OR) | 26.3 [20.8 to NA] — NA is not reached for this entry.
  ER+ and/or PgR+ DR | 14.6 [10.2 to 19.2]
  ER+ and/or PgR+ OR | NA [25.3 to NA] — end number was not reached (NR). not enough data NA is not reached for the confidence interval entry.
  ER-/PgR- DR | 6.2 [4.2 to 10.6]
  ER-/PgR- OR | 18.6 [14.4 to 26.1]
  Adjuvantb Chemotherapy Including Taxane DR | 18.2 [7.2 to 23.6]
  Adjuvantb Chemotherapy Including Taxane OR | 26.1 [17.4 to NA] — NA is not reached for this entry.
  Adjuvantb Chemotherapy Without Taxane DR | 13.2 [10.2 to 15.7]
  Adjuvantb Chemotherapy Without Taxane OR | NA [15.0 to NA] — end number was not reached (NR). not enough data NA is not reached for the confidence interval entry.
  No Previous Adjuvant Chemo DR | 9.0 [4.5 to 19.2]
  No Previous Adjuvant Chemo OR | 26.3 [22.1 to NA] — NA is not reached for this entry.

3. Secondary Outcome: Comparison of Safety and Toxicity
Description: Evaluated using adverse event (AE) information. Detailed AE information is provided in the AE section.
Time Frame: When adverse events occur, up to 30 days after last dose for each subject, up to 3 years from start of study
Measure: Number; unit: subjects
Arm/Group | Docetaxel + Bevacizumab
Number analyzed (Participants) | 76
subjects
  dose reduction of docetaxel for toxicity | 10
  dose delay or interruption | 19
  discontinued docetaxel and continued to receive be | 10
  bevacizumab dose delay or interruption | 24
  patients came off of study because of bevacizumab- | 9

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data collected between 03/2005 and 11/2009. AE reporting period is 4 years 8 months.
Description: Systemic adverse event assessment occurred every 21 days through investigator assessment during treatment period.
Groups:
- Docetaxel and/or Bevacizumab: docetaxel: 75 mg/m2 IV q3 weeks. Bevacizumab: 15mg/kg IV q3 weeks. Subjects continue on dosing until they experience unacceptable toxicity, disease progression, or withdrawal of patient consent.
Arm/Group | Docetaxel and/or Bevacizumab
Serious Adverse Events (participants affected / at risk) | 13/74
Other Adverse Events (participants affected / at risk) | 74/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and/or Bevacizumab (N=74)
Infection (Infections and infestations) | 1
febrile neutropenia (Infections and infestations) | 3
left ventricular dysfunction (Cardiac disorders) | 1
fistula enterovesical (Gastrointestinal disorders) | 1
hemorrhage/bleeding (Vascular disorders) | 2
constipation and hypokalemia (Gastrointestinal disorders) | 1
nausea, vomiting and burning abdominal pain (Gastrointestinal disorders) | 2
speech impairment (Nervous system disorders) | 1
pulmonary embolism (Vascular disorders) | 1
dyspnea, pain (Respiratory, thoracic and mediastinal disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and/or Bevacizumab (N=74)
neutropenia (Blood and lymphatic system disorders) | 25
leukopenia/lymphopenia (Blood and lymphatic system disorders) | 19
febrile neuropenia (Blood and lymphatic system disorders) | 2
anemia (Blood and lymphatic system disorders) | 1
fatigue (General disorders) | 17
fever (General disorders) | 3
insomnia (General disorders) | 3
mucositis/esophagitis/dysphagia (Gastrointestinal disorders) | 6
diarrhea (Gastrointestinal disorders) | 2
anorexia (Gastrointestinal disorders) | 2
nausea/vomiting (Gastrointestinal disorders) | 3
dehydration (Gastrointestinal disorders) | 3
colitis (Gastrointestinal disorders) | 1
infection (Infections and infestations) | 13
pain (General disorders) | 12
hypertension (Cardiac disorders) | 7
thromboembolism (Vascular disorders) | 3
left ventricular dysfunction (Cardiac disorders) | 1
electrolyte abnormality/hyperglycemia (Metabolism and nutrition disorders) | 11
neuropathy (Nervous system disorders) | 2
syncope (Nervous system disorders) | 2
other (Nervous system disorders) | 6
dermatology (Skin and subcutaneous tissue disorders) | 4
dyspnea/hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
mood alteration (Psychiatric disorders) | 6
hemorrhage (Blood and lymphatic system disorders) | 3
epistaxis (Blood and lymphatic system disorders) | 2
hematemesis (Gastrointestinal disorders) | 1
proteinuria (Renal and urinary disorders) | 2
lymphadenopathy (Blood and lymphatic system disorders) | 2

LIMITATIONS AND CAVEATS:
Small sample size and that it was changed from a 2-arm study to a single arm study. This was necessary with public release of E2100 results(improved progression free survival) and subsequent availability of bevacizumab outside of clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No